CLINICAL TRIAL: NCT05692583
Title: Correlation Between EPB Entrapment Test and Ultrasound Wrist Findings in Patients With deQuervain's Disease
Status: Completed | Type: Observational
Sponsor: Velammal Medical College Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Vijayaraja Elangovan, assistant professor in orthopaedics, principal investigator, Velammal Medical College Hospital and Research Institute
Other Study IDs: VMCIEC/27/2022
Record Dates: First submitted 2023-01-08; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: De Quervain Disease
Keywords: de quervain's disease; anatomical variations; EPB entrapment test
MeSH Terms: conditions — De Quervain Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound examination of wrist — musculoskeletal ultrasound examination of affected wrist

SUMMARY:
The goal of this observational study is to learn about the correlation between EPB entrapment test and ultrasound wrist findings in patients with deQuervain's disease The main questions it aims to answer are:

* if correlation exist between EPB entrapment test and ultrasound wrist findings in patients with deQuervain's disease ?
* if the the correlation aid in deciding management of patients with deQuervain's disease Participants will be subjected to
* EPB entrapment test
* ultrasound examination of wrist

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Radial side wrist pain
* Finkelstein test positive
* Failure of non surgical treatment

Exclusion Criteria:

• Patients who underwent Previous surgical release

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all adults >18 years of age with positive Finkelsteins test are included
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
EPB entrapment test | 1 day
  comparing the pain elicited during resisted thumb MCP joint abduction and resisted thumb MCP joint extension
Ultrasound examination of wrist | 1 day
  musculoskeletal ultrasound of affected wrist is done for examining the anatomical variations of first extensor compartment

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasan Rajappa, MS, DNB, Study Director — Sri Ramachandra Institute of Higher Education and Research; Vijayaraja Elangovan, MS, Study Chair — Velammal Medical College Hospital and Research Institute; Gokul Kumar Jeganathan, MBBS, Principal Investigator — Velammal medical college hospital and research
Locations (1):
- Velammal medical college hospital and research institute, Madurai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finkelstein H. STENOSING TENDOVAGINITIS AT THE RADIAL STYLOID PROCESS. JBJS. 1930 Jul;12(3):509-40.
- [Background] E E. Zur Pathogenese der Tendovaginitis stenosans. Bruns Beitrage Z Klin Chir. 1927;0:746-55.
- [Background] GILES KW. Anatomical variations affecting the surgery of de Quervain's disease. J Bone Joint Surg Br. 1960 May;42-B:352-5. doi: 10.1302/0301-620X.42B2.352. No abstract available. PMID 13850049
- [Background] Alexander RD, Catalano LW, Barron OA, Glickel SZ. The extensor pollicis brevis entrapment test in the treatment of de Quervain's disease. J Hand Surg Am. 2002 Sep;27(5):813-6. doi: 10.1053/jhsu.2002.35309. PMID 12239669
- [Background] Lee KH, Kang CN, Lee BG, Jung WS, Kim DY, Lee CH. Ultrasonographic evaluation of the first extensor compartment of the wrist in de Quervain's disease. J Orthop Sci. 2014 Jan;19(1):49-54. doi: 10.1007/s00776-013-0481-3. Epub 2013 Oct 17. PMID 24132793